CLINICAL TRIAL: NCT03390686
Title: A Randomised, Double-blind, Parallel Group, Equivalence, Multicentre Phase III Trial to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity of HD204 to Avastin® in Patients With Metastatic or Recurrent Non-squamous Non-small Cell Lung Cancer
Brief Title: A Trial to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity of HD204 to Avastin® in Advanced Non-squamous Non-small Cell Lung Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAMSON-II
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD204 (Bevacizumab biosimilar) (Experimental): HD204 + Carboplatin/Paclitaxel
  Interventions: Drug: HD204; Drug: Carboplatin; Drug: Paclitaxel
- Avastin (Bevacizumab) (Active Comparator): Avastin® + Carboplatin/Paclitaxel
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg IV every 3 weeks on Day 1
  Other Names: Avastin
  Arms: Avastin (Bevacizumab)
Drug: HD204 — 15 mg/kg IV every 3 weeks on Day 1
  Other Names: Bevacizumab
  Arms: HD204 (Bevacizumab biosimilar)
Drug: Carboplatin — Carboplatin AUC 6 IV every 3 weeks on Day 1 for 4-6 cycles
Drug: Paclitaxel — Paclitaxel 200 mg/m2 IV every 3 weeks on Day 1 for 4-6 cycles
  Other Names: Taxol

SUMMARY:
In the SAMSON-2 study, the proposed biosimilar HD204 will be compared to its reference product EU-licensed Avastin®. The aim of the study is to demonstrate equivalence of HD204 and EU-licensed Avastin® in terms of efficacy, safety, pharmacokinetics and immunogenicity.

DETAILED DESCRIPTION:
This is a randomised, double-blind, parallel group, equivalence, multicentre Phase III study in patients with metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC).

Standard efficacy parameters, safety profiles, pharmacokinetics and immunogenicity will be compared between HD204 and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* ECOG performance status of 0-1
* Histologically-confirmed metastatic or recurrent non-squamous non-small cell lung cancer
* At least one measurable lesion according to RECIST v1.1.
* Able to receive bevacizumab, carboplatin and paclitaxel based on adequate laboratory and clinical parameters

Exclusion Criteria:

* Diagnosis of small cell carcinoma of the lung or squamous cell carcinoma
* Sensitizing EGFR mutations or ALK rearrangements
* Increased risk of bleeding determined by investigator based on radiographic / clinical findings
* History of systemic chemotherapy administered in the first-line setting for metastatic or recurrent disease of NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Week 18 | 18 weeks from randomization
  Percent patients within each treatment group who achieved complete response (CR) or partial response (PR) by the time of the Week 18 efficacy analysis in accordance with the RECIST 1.1. as assessed by CIR.

SECONDARY OUTCOMES:
ORR at Week 6 | 6 weeks from randomization
  Response at Week 6 will be evaluated by CIR to show the pattern of response
ORR at Week 12 | 12 weeks from randomization
  Response at Week 12 will be evaluated by CIR to show the pattern of response
ORR at Week 18 adjusted on dose intensity | 18 weeks from randomization
  To compare ORR at Week 18 adjusted on dose intensity between treatment groups
Duration of Response | from documented tumour response until disease progression up to 12 months from randomisation
  DoR in subjects with response from documented tumour response until disease progression up to 12 months from randomisation of the last subject
Progression Free Survival | From the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
  PFS from the date of randomisation to the date of disease progression or death up to 12 months from randomisation
Overall Survival (OS) | From the date of randomisation to the date of death up to 12 months from randomisation
  OS defined as the time from Day 1 of therapy until death from any cause
Change in tumour burden from baseline | Up to 52 weeks from baseline
  Measured by the sum of longest diameters (SLD) of the target lesions
Incidence of Treatment-related Adverse Events using CTCAE v5.0 | From signing the ICF until 1 month after the last administration of treatment, i.e., up to 52 weeks
  After the end of treatment (EOT) visit, SAEs should be reported to the Sponsor if the Investigator becomes aware of them.
Anti-Drug Antibodies (Immunogenicity) | Up to 52 weeks (at Baseline; end of Cycle 4 [pre-dose in cycle 5]; end of Cycle 7 [pre-dose in cycle 8]; and at EOT)
  Incidence of anti-drug (bevacizumab) antibodies (ADA)
Neutralizing Antibodies (Immunogenicity) | Up to 52 weeks (at Baseline; end of Cycle 4 [predose in cycle 5]; end of Cycle 7 [predose in cycle 8]; and at EOT)
  Incidence of anti-drug (bevacizumab) antibodies (ADA) - neutralizing antibodies (NAb)
Trough Level [Ctrough] (Pharmacokinetics) | Up to 52 weeks (end of Cycle 1 [predose of Cycle 2], end of Cycle 3 [predose of Cycle 4], end of Cycle 5 [predose of Cycle 6] and EOT)
  Concentration observed 19 to 23 days after study drug administration
Maximum Plasma Concentration [Cmax] (Pharmacokinetics) | Up to 21 weeks (Cycle 2 ,4 and 6. Each cycle is 21 days.)
  Cmax at selected cycles
Area under the concentration-time curve from 0 hr to time t [AUC0-t] (Pharmacokinetics) | Up to 21 weeks (Cycle 2 ,4 and 6. Each cycle is 21 days.)
  AUC0-t at selected cycles

CONTACTS AND LOCATIONS:
Locations (18):
- Alexandrov Cancer Center, Minsk, Minsk City, Belarus
- MHAT "Dr. Tota Venkova", AD, Gabrovo, Bulgaria
- CHC Osijek, Osijek, Osijecko-baranjska, Croatia
- Georgia (2):
  - LTD "High Technology Hospital Medcenter", Batumi
  - Institute of Clinical Oncology, Tbilisi
- Interbalkan Hospital, Thessaloniki, Asklipiou 10, Greece
- Tudogyogyintezet Torokbalint, Törökbálint, Hungary
- HCG Manavata Cancer Centre, Nashik, Maharashtra, India
- Riga East University Hospital Latvian Oncology centre, Riga, Latvia
- HRPZ II, Kota Bharu, Kelantan, Malaysia
- Asian Hospital and Medical Center, City of Muntinlupa, Philippines
- Magodend Szpital Elblaska, Warsaw, Poland
- MEDSI, Moscow, Otradnoye, Russia
- IPD of Vojvodina, Kamenitz, Serbia
- Nemocnica na okraji mesta, n.o., Partizánske, Slovakia
- Maharaj Nakorn Chiang Mai, Chiang Mai, Muang, Thailand
- Acibadem Adana Hospital, Adana, Turkey (Türkiye)
- Oncology Dispensary, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided